CLINICAL TRIAL: NCT00007020
Title: Investigation in the Pathogenesis of Liver Disease in Patients With Inborn Errors of Bile Acid Metabolism
Brief Title: Compassionate Treatment of Patients With Inborn Errors of Bile Acid Metabolism With Cholic Acid
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAC-91-10-10; CCHMC-91-10-10 (Other: Cincinnati Children's Hospital Medical Center); NCRR-M01RR08084-0009 (Other: National Center For Research Resources (NCRR))
Record Dates: First submitted 2000-12-06; First posted 2000-12-07 (Estimated); Results first posted 2020-07-15 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Infantile Refsum's Disease; Zellweger Syndrome; Adrenoleukodystrophy; Peroxisomal Disorders; Cholestasis
MeSH Terms: conditions — Refsum Disease, Infantile; Zellweger Syndrome; Adrenoleukodystrophy; Peroxisomal Disorders; Cholestasis | interventions — Cholic Acids; Cholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cholic Acid (Other)
  Interventions: Drug: Cholic Acids

INTERVENTIONS:
Drug: Cholic Acids — 10-15 mg/kg body weight/day taken orally.
  Other Names: Cholic; Cholic Acid; Cholic Acid Capsules

SUMMARY:
OBJECTIVES:

I. To Evaluate the therapeutic efficacy of cholic acid during provision of compassionate treatment to patients with identified inborn errors of bile acid synthesis and metabolism

II. To assess the safety and tolerability of cholic acid

DETAILED DESCRIPTION:
Investigational Plan:

A Phase III, open label, single arm, nonrandomized, non-comparative, compassionate treatment study of cholic acid in the treatment of defects of bile acid metabolism.

The study was begun with a single study site at Cincinnati Children's Hospital Medical Center (CCHMC), but in 2005 was expanded so that compassionate treatment could be provided to additional patients who had been identified with inborn errors of bile metabolism through the center's screening/diagnostic program.

Patients who were screened were contacted and evaluated with respect to the inclusion/exclusion criteria. Signed informed consent by the patient and/or parents/legal guardian was obtained as soon as it is confirmed that the patient met inclusion/exclusion criteria and the parents/guardian would agree for the child to participate in the study.

The primary interventions for the study were:

1. Administration of study drug.
2. Collection of baseline physical exam, vital signs, blood and urine samples for laboratory tests.
3. Collection of periodic physical exam, vital signs, blood and urine samples for laboratory tests during the period of administration of the study drug.
4. Collection of any adverse event information.

Time and Events Schedule:

Baseline:

1. Confirm eligibility
2. Obtain written informed consent from patient and/or parents/legal guardian
3. Collect demographic data and disease and medication history, including family history

   Baseline and Ongoing:
4. Obtain body weight
5. Record adverse events
6. Obtain blood and urine samples for laboratory tests
7. Initiate study drug therapy & monitor study drug therapy and adjust dose as needed

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Clinical or biochemical evidence of liver disease, unexplained fat-soluble vitamin malabsorption, or peroxisomal dysfunction that compromises bile acid biosynthesis

Inclusion criteria for enrollment were:

* Infants < age 3 months
* Children presenting for evaluation of cholestasis defined as a conjugated bilirubin > 2mg/dl or increased serum bile acids
* Older subjects of any age with cholestatic liver disease if urine screens suggested that they had inborn errors of bile acid metabolism
* Confirmation of a diagnosis of an inborn error of bile acid synthesis based upon urine analysis by FAB-MS to determine whether specific abnormalities in bile acid synthesis are indicated
* The patient and/or parent/legal guardian must have signed the written informed consent document before study start.
* The patient must be willing and able to comply with all study assessments and procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 1992-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Heubi, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Kenneth Setchell, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Heubi JE, Bove KE, Setchell KDR. Oral Cholic Acid Is Efficacious and Well Tolerated in Patients With Bile Acid Synthesis and Zellweger Spectrum Disorders. J Pediatr Gastroenterol Nutr. 2017 Sep;65(3):321-326. doi: 10.1097/MPG.0000000000001657. PMID 28644367

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 85 patients were enrolled.
Pre-assignment Details: Of the patients diagnosed with a defect in bile acid synthesis during routine diagnostic procedures at the Cincinnati Children's Hospital Medical Center (CCHMC) Mass Spectrometry Laboratory, 85 patients were invited to participate in the study.
Groups:
- Cholic Acid: Cholic acid capsules, each containing 250 mg of cholic acid, or a liquid preparation of 15 mg/mL cholic acid, to be administered orally in a dose of 15 mg/kg body weight/day.
Period: Overall Study
Arm/Group | Cholic Acid
Started | 85
Completed | 41
Not Completed | 44
Not completed — Death | 16
Not completed — Lost to Follow-up | 13
Not completed — Pt withdrawn (worsening cholestasis) | 1
Not completed — Pt withdrawn (liver transplant) | 4
Not completed — Pt cared for by outside physician | 4
Not completed — No evidence of treatment | 6

BASELINE CHARACTERISTICS:
Groups:
- Cholic Acid: All patients entered into the study
Arm/Group | Cholic Acid
Number analyzed (Participants) | 85
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Continuous age data were not available for 8 out of 85 patients.
  years
    number analyzed (Participants) | 77
    (all) | 3 (4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Information on gender was not recorded for 4 patients.
  Participants
    number analyzed (Participants) | 81
    Female | 31
    Male | 50
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 85

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Excretion of Atypical Bile Acids in Urine by Category
Description: Patients with excretion of atypical bile acids in urine by category, from worst status before treatment (baseline, BL) to best status on treatment (OT)
Time Frame: Baseline, then every 1, 3, or 6 months (depending on protocol version) for an average of 2.8 years
Population: Patients treated and with at least 1 pre-treatment and 1 post-treatment assessment
Measure: Count of Participants; unit: Participants
Groups:
- Cholic Acid: Patients treated
Arm/Group | Cholic Acid
Number analyzed (Participants) | 70
Participants
  Baseline, no atypical bile acid excretion | 10
  On treatment, no atypical bile acid excretion | 51
  Baseline, slight atypical bile acid excretion | 11
  On treatment, slight atypical bile acid excretion | 9
  Baseline, significant atypical bile acid excretion | 16
  OT, significant atypical bile acid excretion | 4
  Baseline, marked atypical bile acid excretion | 33
  On treatment, marked atypical bile acid excretion | 6

2. Secondary Outcome: Change in Liver Function Tests (LFTs) Measured in Serum
Description: Patients with elevations of liver function tests (alanine transaminase [ALT], aspartate transaminase [AST]) measured as multiples of the upper limit of normal (ULN) at baseline (worst value) and on treatment (best value)
Time Frame: Baseline, then every 1, 3, or 6 months (depending on protocol version) for an average of 2.8 years
Population: Patients treated and with at least 1 pre-treatment and 1 post-Treatment assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Cholic Acid
Number analyzed (Participants) | 70
Participants
  Baseline, ALT <ULN | 14
  On treatment, ALT <ULN | 49
  Baseline, ULN ≤ ALT <2 x ULN | 16
  On treatment, ULN ≤ ALT <2 x ULN | 13
  Baseline, 2 ULN ≤ ALT <3 x ULN | 8
  On treatment, 2 ULN ≤ ALT <3 x ULN | 2
  Baseline, ALT ≥3 x ULN | 29
  On treatment, ALT ≥3 x ULN | 3
  Baseline, AST <ULN | 9
  On treatment, AST <ULN | 38
  Baseline, ULN ≤ AST <2 x ULN | 14
  On treatment, ULN ≤ AST <2 x ULN | 15
  Baseline, 2 ULN ≤ AST <3 x ULN | 7
  On treatment, 2 ULN ≤ AST <3 x ULN | 4
  Baseline, AST ≥3 x ULN | 35
  On treatment, AST ≥3 x ULN | 9

3. Secondary Outcome: Liver Histology
Description: Patients (number, percentage) with pathological findings for qualitative (the presence of inflammation, fibrosis, necrosis, giant cells and cholestasis) and quantitative (the degrees of the aforementioned histologic features) liver histopathology at baseline (BL) and on treatment (OT).
Time Frame: At baseline (if no historical data were available) and between 1 and 6 months following treatment start.
Population: All patients entered into the study
Measure: Count of Participants; unit: Participants
Arm/Group | Cholic Acid
Number analyzed (Participants) | 85
Participants
  Periportal inflammation at BL, qualitative | 19
  Periportal inflammation OT, qualitative | 16
  Lobular inflammation at BL, qualitative | 5
  Lobular inflammation OT, qualitative | 4
  Inflammation (not spec.) at BL, qualitative | 3
  Inflammation (not spec.) OT, qualitative | 0
  Bridging fibrosis at BL, qualitative | 25
  Bridging fibrosis OT, qualitative | 31
  Fibrosis (not specified) at BL, qualitative | 6
  Fibrosis (not specified) OT, qualitative | 6
  Cholestasis at BL, qualitative | 20
  Cholestasis OT, qualitative | 10
  Giant cells at BL, qualitative | 18
  Giant cells OT, qualitative | 12
  Necrosis at BL, qualitative | 14
  Necrosis OT, qualitative | 2
  Periportal inflammation at BL, quantitative | 18
  Periportal inflammation OT, quantitative | 15
  Lobular inflammation at BL, quantitative | 5
  Lobular inflammation OT, quantitative | 4
  Inflammation (not specified) at BL, quantitative | 3
  Inflammation (not specified) OT, quantitative | 0
  Bridging fibrosis at baseline, quantitative | 22
  Bridging fibrosis OT, quantitative | 27
  Fibrosis (not specified) at BL, quantitative | 3
  Fibrosis (not specified) OT, quantitative | 5
  Cholestasis at BL, quantitative | 15
  Cholestasis OT, quantitative | 7
  Giant cells at BL, quantitative | 13
  Giant cells OT, quantitative | 9
  Necrosis at BL, quantitative | 13
  Necrosis OT, quantitative | 2

4. Secondary Outcome: Height and Weight
Description: Change in height/weight percentiles from baseline (worst value) to the best on-treatment value, based on CDC (Centres for Disease Control and Prevention, US) growth chart percentiles
Time Frame: Baseline, then every 1, 3, or 6 months (depending on protocol version) for an average of 2.8 years
Population: Patients treated and with at least 1 pre-treatment and 1 post-treatment assessment
Measure: Mean (Standard Error); unit: Percentile
Arm/Group | Cholic Acid
Number analyzed (Participants) | 70
Percentile
  Height percentile, baseline | 30.1 (5.5)
  Height percentile, on treatment | 44.0 (6.1)
  Weight percentile, baseline | 21.3 (3.7)
  Weight percentile, on treatment | 42.3 (4.8)

5. Secondary Outcome: Adverse Events
Description: Number of patients with any adverse event
Time Frame: Baseline, then every 1, 3, or 6 months (depending on protocol version) for an average of 2.8 years
Population: Patients entered into the study and treated
Measure: Count of Participants; unit: Participants
Groups:
- Cholic Acid: All patients entered into the study and treated
Arm/Group | Cholic Acid
Number analyzed (Participants) | 79
Participants
  Patients at risk | 79
  Patients with any AE | 38

6. Other Pre Specified Outcome: Change in Bilirubin Measured in Serum
Description: Bilirubin concentration in serum at baseline and on treatment
Time Frame: Baseline and on treatment (every 1, 3, or 6 months, depending on protocol version, for an average of 2.8 years)
Population: All available bilirubin laboratory data are collected then grouped by bilirubin test type and collection time points (baseline vs. on treatment). Not all participant had available data, and each participant may have more than one type of bilirubin collected at a time point, and may have multiple on-treatment collections.
Measure: Mean (Standard Deviation); unit: mg/dL
Units Other Than Participants: Number of Test Results
Arm/Group | Cholic Acid
Number analyzed (Participants) | 60
Number analyzed (Number of Test Results) | 689
mg/dL
  Baseline, bilirubin: number analyzed (Participants) | 1
  Baseline, bilirubin: number analyzed (Number of Test Results) | 1
  Baseline, bilirubin | 0.3
  On treatment, bilirubin: number analyzed (Participants) | 6
  On treatment, bilirubin: number analyzed (Number of Test Results) | 15
  On treatment, bilirubin | 0.6 (0.5)
  Baseline, direct bilirubin: number analyzed (Participants) | 31
  Baseline, direct bilirubin: number analyzed (Number of Test Results) | 82
  Baseline, direct bilirubin | 2.2 (5.6)
  On treatment, direct bilirubin: number analyzed (Participants) | 44
  On treatment, direct bilirubin: number analyzed (Number of Test Results) | 195
  On treatment, direct bilirubin | 0.5 (1.8)
  Baseline, indirect bilirubin: number analyzed (Participants) | 5
  Baseline, indirect bilirubin: number analyzed (Number of Test Results) | 5
  Baseline, indirect bilirubin | 0.5 (0.9)
  On treatment, indirect bilirubin: number analyzed (Participants) | 7
  On treatment, indirect bilirubin: number analyzed (Number of Test Results) | 17
  On treatment, indirect bilirubin | 0.2 (0.2)
  Baseline, total bilirubin: number analyzed (Participants) | 28
  Baseline, total bilirubin: number analyzed (Number of Test Results) | 86
  Baseline, total bilirubin | 2.8 (10.6)
  On treatment, total bilirubin: number analyzed (Participants) | 48
  On treatment, total bilirubin: number analyzed (Number of Test Results) | 288
  On treatment, total bilirubin | 1.5 (5.2)

ADVERSE EVENTS:
Time Frame: Baseline, then every 1, 3, or 6 months (depending on protocol version) for an average of 2.8 years
Groups:
- Cholic Acid: All patients entered into the study and treated with Cholic Acid. 85 patients enrolled in the study and 79 received treatment (safety set).
Arm/Group | Cholic Acid
All-Cause Mortality (participants affected / at risk) | 13/79
Serious Adverse Events (participants affected / at risk) | 20/79
Other Adverse Events (participants affected / at risk) | 35/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cholic Acid (N=79)
Nutritional condition abnormal (Investigations) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Disease progression (General disorders) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (2)
Infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Rotavirus infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cholic Acid (N=79)
Disease progression (General disorders) | 1 (1)
Injection site inflammation (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Pyrexia (General disorders) | 7 (7)
Hallucination (Psychiatric disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Ovarian failure (Reproductive system and breast disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 4 (6)
Amino acid level increased (Investigations) | 1 (1)
Occult blood (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Convulsion (Nervous system disorders) | 4 (6)
Hypotonia (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Enteritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
Vitamin E deficiency (Metabolism and nutrition disorders) | 2 (2)
Bronchopneumonia (Infections and infestations) | 2 (2)
Ear infection (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (2)
Otitis media (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (5)
Varicella (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
CAC-91-10-10 includes data from patients enrolled from 1992-2009. The study end date was arbitrarily chosen as data cut-off point; the disease requires life-long treatment, no final study visit was done. Many patients continued onto study CAC-002-01

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No